CLINICAL TRIAL: NCT03757676
Title: Effects of Playing Pokemon Go on Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: University of Southern California (Other)
Responsible Party: Principal Investigator, Noe Crespo, Assistant Professor, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HS-2017-0235
Record Dates: First submitted 2018-11-27; First posted 2018-11-29 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Physical Activity
Keywords: Physical Activity; Mobile Games
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned into one of three experimental groups: a control group and two play groups. The two play groups consisted of a group that was asked to play Pokémon Go ad libitum (at will play) and the other group was asked to achieve a specific level within the game during the study period (goal oriented play). Participants were measured for baseline physical activity levels (2 weeks) followed by randomization to one of the three groups. The intervention period lasted 4 weeks. All participants completed a brief questionnaire and were measured for height and weight, and daily physical activity levels using a FitBit accelerometer. Locations of where individual engaged in physical activity were recorded using a GPS tracking application. During the 5th week of the study period, participants completed five (5) short surveys per day using Ecological Momentary Assessment (EMA) software to assess level of play and engagement of play.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No Play (Experimental): This 'no play' group functioned as the control group.
  Interventions: Behavioral: No Play
- At Will Play (Experimental): This group functioned as 1 of the 2 play groups.
  Interventions: Behavioral: At Will Play
- Goal Oriented Play (Experimental): This group functioned as 1 of the 2 play groups.
  Interventions: Behavioral: Goal Oriented Play

INTERVENTIONS:
Behavioral: No Play — Participants in this group were asked not to download or play Pokémon Go during the study period and were asked to simply continue with their normal daily activities. Participants were asked to wear the Fitbit device and use the GPS app on their mobile phones during the 6-week study period. Starting the fifth week, participants were prompted to complete five (5) brief daily surveys on their phones via the EMA app.
  Arms: No Play
Behavioral: At Will Play — Participants in this group were asked to download Pokémon Go and play for at least 30 minutes initially, then play as much or as little as desired during the 4 week intervention period, with no specific instruction or goals for play. Participants were asked to wear the Fitbit device and use the GPS app on their mobile phones during the 6-week study period. Starting the fifth week, participants were prompted to complete five (5) brief daily surveys on their phones via the EMA app.
  Arms: At Will Play
Behavioral: Goal Oriented Play — Participants in this group were asked to download and play Pokémon Go and achieve a minimum player level of 20 within the game during the study period. They were given materials that described game features and functions to show them how to play the game. There were no restrictions on which features to pursue within the game to achieve this goal nor on how long or how frequent their play sessions should be. Upon reaching their goal (Level 20), participants were encouraged to continue to play as much or as little as they desired. Participants were asked to wear the Fitbit device and use the GPS app on their mobile phones during the 6-week study period. Starting the fifth week, participants were prompted to complete five (5) brief daily surveys on their phones via the EMA app.
  Arms: Goal Oriented Play

SUMMARY:
The purpose of this study was to test the feasibility and preliminary efficacy of playing Pokémon Go to increase daily steps among young adults. The study also aimed to assess people's experience playing the game, identify specific features of the game that users like/dislike, and explore game features that may promote overall well-being.

DETAILED DESCRIPTION:
Study participants were 30 undergraduate students from a State university in California who were 18 years or older, enrolled full-time, non-Pokémon Go players, and were able to walk leisurely. Daily steps were measured for 6 consecutive weeks via the Fitbit Flex 2. Habitual activity was first measured during the first two-weeks. After the 2-week baseline assessment of physical activity and GPS travel patterns, participants were randomized to one of three study conditions for the remaining 4 weeks: (1) "No Play," (2) "Play At Will," or (3) "Goal Oriented Play". The 4-week intervention period was followed by a post-study interview completed within one week from the end of the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled as a full-time undergraduate or graduate student at participating University
* Willingness to be randomized to one of the three study conditions
* Never played or a Novice Player of Pokemon Go (Cannot have previously exceeded Level 5)
* Not currently meeting physical activity guidelines for adults (i.e., 150 minutes per week of moderate-intensity aerobic activity and/or 75 minutes per week of vigorous-intensity aerobic activity). Assessed via the GPAQ questionnaire.

Exclusion Criteria:

- Unable to leisurely walk for 30 minutes consecutively

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2018-03-22 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Steps per day | Six weeks
  Steps per day measured via the Fitbit

CONTACTS AND LOCATIONS:
Overall Officials: Noe C Crespo, PhD, Principal Investigator — San Diego State University
Locations (1):
- Institute for Behavioral and Community Health, San Diego, California, United States